CLINICAL TRIAL: NCT02204163
Title: A Phase III, Multi-center, Randomized, Comparative, Parallel, Open Study to Assess the Efficacy and Safety After Treatment of Eutropin® Inj. Compared to Genotropin® in Infants/Toddlers With Prader-Willi Syndrome
Brief Title: Study to Assess the Efficacy and Safety of Eutropin in Prader-Willi Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-HGCL007
Record Dates: First submitted 2014-07-25; First posted 2014-07-30 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Human Growth Hormone

ARMS (2):
- Eutropin (Experimental): Eutropin 0.24mg/kg/week
  Interventions: Drug: Eutropin
- Genotropin (Active Comparator): Genotropin 0.24mg/kg/week
  Interventions: Drug: Genotropin

INTERVENTIONS:
Drug: Eutropin
  Arms: Eutropin
Drug: Genotropin
  Arms: Genotropin

SUMMARY:
Evaluate the efficacy and safety after treatment of Eutropin® inj. compared to Genotropin® in infants/toddlers with Prader-Willi syndrome

ELIGIBILITY:
* Inclusion Criteria:

  1. Pediatric patients with PWS confirmed by methylation PCR genetic testing
  2. Prepubertal pediatric patients (Tanner's Pubertal stage I) at screening
  3. Pediatric patients who have never been treated with hGH prior to screening, or who had been treated with hGH for less than 6 months if they had a treatment history, and whose last administration was made 6 months prior to screening
  4. Pediatric patients with normal thyroid function at screening (Those with normal function through a hormonal therapy were allowable.)
  5. Pediatric patients whose parents or LARs signed the informed consent form in writing after receiving the explanation about the purpose, method, effects, etc. of the clinical study, and who also signed the informed consent form in writing if they are capable of reading and understanding writing.
* Exclusion Criteria:

  1. Pediatric patients who are accompanied by other causes for growth retardation as follows except for PWS at screening

     : Chronic renal failure (including the case in which renal transplantation has been undergone), Silver-Russell syndrome, Turner's syndrome, Seckel syndrome, Down's syndrome, Noonan syndrome, Cushing's syndrome, congenital infections, psychiatric disorders, chronic debilitating diseases, etc.
  2. Pediatric patients with malignancy or a history of malignancy at screening
  3. Pediatric patients with severe respiratory disturbance, or sleep apnoea or a history of respiratory infections with an unknown cause at screening. However, those whose condition had been confirmed to be eligible to participate in the clinical study on investigator's judgment were allowed to participae in the study.
  4. Pediatric patients with impaired fasting glucose, diabetes, and diabetic retinopathy at screening
  5. Pediatric patients whose epiphyses are closed with a growth rate of ≤1 cm/year at screening
  6. Pediatric patients who are being administered any drug that may have an effect on the secretion and actions of hGH (estrogen, androgen, anabolic steroids, corticosteroids, GnRH analogs, thyroxine, aromatase inhibitors, etc.) or anticonvulsants and cyclosporin at screening, and have been administered any of them for a long period of time within 6 months prior to screening (However, those who have been administered a thyroxine preparation for ≥4 weeks on a stable dose [allowable in case the investigator determines the dose is stable even though it is changeable based upon the weight of the pediatric patient] were allowed to participate in the clinical study.)
  7. Pediatric patients who are being administered any drug (e.g. methylphenidate) for treatment of hyperactivity disorders including attention deficit hyperactivity disorder (ADHD) at screening
  8. Pediatric patients who are hypersensitive to somatropin or any excipient of the investigational product (cresol or glycerol) or who have a relevant history of hypersensitivity
  9. Pediatric patients who have participated in any other clinical studies after enrolled in this study or who had participated in any other clinical studies within 3 months prior to enrollment in this clinical study
  10. Pediatric patients in whom this clinical study is considered to be difficult to be conducted for any other reasons on investigator's judgment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in height SDS (Standard Deviation Score) | baseline and 52 weeks
Change from baseline in Lean body mass (g) | baseline and 52 weeks
Change from baseline in Percent body fat (%) | baseline and 52 weeks

SECONDARY OUTCOMES:
Change from baseline in height velocity (cm/year) | baseline, 16, 28 and 52 weeks
Change from baseline in head circumference (cm) | baseline, 16, 28 and 52 weeks
Change from baseline in cognitive development (score) by Bayley Scale | baseline, 28 and 52 weeks
Change from baseline in motor development (score) by Bayley Scale | baseline, 28 and 52 weeks
Change from baseline in weight SDS | baseline 16, 28 and 52 weeks
Change from baseline in BMI (kg/m2) (Body Mass Index) | baseline, 16, 28 and 52 weeks
Change from baseline in Bone age (month) | baseline and 52 weeks
Change from baseline in Bone mineral density (g/cm) | baseline and 52 weeks
Change from baseline in height (cm) | baseline, 16, 28 and 52 weeks
Change from baseline in height SDS | baseline, 16 and 28 weeks
Change from baseline in IGF-1 (ng/mL) and IGF-1 SDS | baseline, 28, and 52 weeks
Change from baseline in IGFBP-3 (ng/mL) and IGFBP-3 SDS | baseline, 28, and 52 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Yang A, Choi JH, Sohn YB, Eom Y, Lee J, Yoo HW, Jin DK. Effects of recombinant human growth hormone treatment on growth, body composition, and safety in infants or toddlers with Prader-Willi syndrome: a randomized, active-controlled trial. Orphanet J Rare Dis. 2019 Sep 11;14(1):216. doi: 10.1186/s13023-019-1195-1. PMID 31511031